CLINICAL TRIAL: NCT06859099
Title: Long-term Extension Study to Evaluate the Safety and Efficacy of Riliprubart (SAR445088) in Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Long-term Safety and Efficacy Study of Riliprubart in Participants With CIDP
Acronym: LTS
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17261; U1111-1311-1432 (Other: WHO ICTRP); 2024-517032-22-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Polyneuropathy, Inflammatory Demyelinating, Chronic
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- riliprubart (Experimental): Participants receive subcutaneous injection with a riliprubart prefilled pen (PFP)
  Interventions: Drug: Riliprubart Prefilled Pen (PFP)

INTERVENTIONS:
Drug: Riliprubart Prefilled Pen (PFP) — Pharmaceutical form: Solution Route of administration: Subcutaneous injection
  Other Names: SAR445088

SUMMARY:
This study is a Phase 3 extension, global, multicenter open-label study. The purpose of this study is to evaluate long-term safety and efficacy of riliprubart in adult participants with chronic inflammatory demyelinating polyneuropathy (CIDP) who have completed Part B in 1 of 3 parent studies (PDY16744, EFC17236, or EFC18156) and wish to continue treatment with riliprubart. Up to approximately 300 participants will be enrolled to continue receiving treatment with riliprubart. The duration of participation for each participant will be up to approximately 4 years, including posttreatment follow-up. The treatment duration will be up to approximately 3 years. A participant who discontinues riliprubart treatment at any time during the study will be followed for safety for a minimum of 55 weeks after the last dose of riliprubart received.

DETAILED DESCRIPTION:
This is a single-arm study. All participants transitioning to Study LTS17261 will receive riliprubart weekly for up to 3 years, or until commercialization of riliprubart for the treatment of CIDP or termination of the riliprubart clinical development program for the treatment of CIDP, or the local availability of other options for long-term treatment with riliprubart, whichever comes first.

The total number of study visits will be 12.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participants with chronic inflammatory demyelinating polyneuropathy (CIDP) currently receiving riliprubart who completed treatment in Part B of Study PDY16744, Study EFC17236, or Study EFC18156. (Participants receiving riliprubart in Part C of PDY16744 are eligible after completing the Part C End of Treatment visit.)
2. All participants must agree to use contraception methods during and after the study as required. Contraceptive use by men and women participating in the study should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
3. Participant must be capable of giving signed informed consent as described in Appendix 1 of the protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Pregnancy, defined as a positive result of a highly sensitive urine or serum pregnancy test, or lactation
2. Clinical diagnosis of systemic lupus erythematosus (SLE)
3. History of any hypersensitivity to riliprubart or any of its components, or severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibody
4. Any country-related specific regulation that would prevent the participant from entering the study
5. Accommodation in an institution because of regulatory or legal order; for instance, a prisoner or participant who is legally institutionalized
6. Unsuitability for participation as judged by the Investigator, whatever the reason, including: medical or clinical condition, potential risk of participant noncompliance with study procedures, or any other clinically significant change in the participants' medical condition

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-10-03 (Estimated); Study Completion 2029-10-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants having any AEs, SAEs, adverse events leading to treatment discontinuation, AESIs, and potentially clinically significant abnormalities (PCSAs) in safety laboratory tests, ECGs, and vital signs during the study period | Up to End of Study (approx. 4 years)
  adverse events: AEs, serious adverse events: SAEs, adverse events of special interest: AESIs, electrocardiograms: ECGs

SECONDARY OUTCOMES:
Percentage of participants relapse-free since the first dose of riliprubart in the parent study (PDY16744, EFC17236, or EFC18156) | From first dose of riliprubart in parent study to end of treatment (up to approx. 7 years)
  To estimate the relapse-free rate, time to first relapse, defined as time from first dose of riliprubart in the parent study to the first relapse since riliprubart initiation, will be derived for each participant. Relapse since riliprubart initiation is defined as increase of 1 point or more in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score relative to the visit for the first dose of riliprubart in the parent study.
Percentage of participants experiencing improvement from baseline | From Baseline to 3 years
  Improvement is defined as a decrease of 1 point or more in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score relative to baseline of the current study, Study LTS17261
Change from baseline in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score over time | From Baseline to 3 years
Change from baseline in Inflammatory Rasch-built Overall Disability Scale (I-RODS) over time | From Baseline to 3 years
Change from baseline in grip strength (kilopascals; dominant hand) over time | From Baseline to 3 years
Change from baseline in Medical Research Council-Sum Score (MRC-SS) for muscle strength over time | From Baseline to 3 years

CONTACTS AND LOCATIONS:
Locations (36):
- United States (2):
  - Alabama Neurology Associates- Site Number : 8400019, Homewood, Alabama
  - University of Kansas Medical Center- Site Number : 8400010, Kansas City, Kansas
- Canada (2):
  - Investigational Site Number : 1240001, Gatineau, Quebec
  - Investigational Site Number : 1240002, Québec, Quebec
- Chile (2):
  - Investigational Site Number : 1520003, Lo Barnechea, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- China (6):
  - Investigational Site Number : 1560013, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560011, Chengdu
  - Investigational Site Number : 1560002, Fuzhou
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560003, Wuhan
- Investigational Site Number : 2030004, Brno, Czechia
- Investigational Site Number : 2080002, Aarhus, Denmark
- France (5):
  - Investigational Site Number : 2500007, Bordeaux
  - Investigational Site Number : 2500001, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500005, Montpellier
  - Investigational Site Number : 2500004, Paris
- Germany (2):
  - Investigational Site Number : 2760002, Göttingen
  - Investigational Site Number : 2760004, Tübingen
- Italy (6):
  - Investigational Site Number : 3800003, Genoa, Genova
  - Investigational Site Number : 3800001, Milan, Milano
  - Investigational Site Number : 3800004, Rozzano, Milano
  - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800005, Pavia
  - Investigational Site Number : 3800007, Pisa
- Investigational Site Number : 5280001, Amsterdam, Netherlands
- Investigational Site Number : 6160001, Lublin, Lublin Voivodeship, Poland
- Investigational Site Number : 6880001, Belgrade, Serbia
- Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi, South Korea
- Spain (4):
  - Investigational Site Number : 7240004, Majadahonda, Madrid
  - Investigational Site Number : 7240002, Barcelona
  - Investigational Site Number : 7240001, Barcelona
  - Investigational Site Number : 7240003, Valencia
- Investigational Site Number : 7520001, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17261 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26640&tenant=MT_SNY_9011